CLINICAL TRIAL: NCT04663282
Title: Evaluation of the Efficacy and Safety of INS068 Injection and Insulin Degludec Subcutaneous Injection Once Daily in Subjects With Type 2 Diabetes Mellitus Not Adequately Controlled With One or Two Oral Antidiabetics (A Randomized, Open-Label, Two-Arm, Treat-to-Target, Parallel Controlled Trial)
Brief Title: A Trial of INS068 in Patients With Type 2 Diabetes Not Adequately Controlled With One or Two Oral Antidiabetics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INS068-201
Record Dates: First submitted 2020-12-02; First posted 2020-12-10 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Intervention Model Description: INS068 campared with Insulin degludec, both in Combination with One or Two Oral Antidiabetics
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- INS068 (Experimental): Intervention: Drug: INS068 injection
  Interventions: Drug: INS068 injection
- IDeg (Active Comparator): Intervention: Drug: insulin Degludec
  Interventions: Drug: Insulin Degludec

INTERVENTIONS:
Drug: INS068 injection — INS068 injected subcutaneously once daily. Treat-to-target dose titration during the trial
  Arms: INS068
Drug: Insulin Degludec — Insulin Degludec injected subcutaneously once daily. Treat-to-target dose titration during the trial
  Arms: IDeg

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of IND068 once daily (QD) in subjects with type 2 diabetes not adequately controlled with one or two oral antidiabetics compared to insulin degludec QD for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that will not have been performed during normal management of the subject.)
* Age is 18-75 years
* Diagnosed with Type 2 diabetes (according to the diagnosis criteria applicable locally) for at least 3 months
* Treatment with one or two oral anti-diabetic drug (OADs): metformin at astable daily dose of ≥ 1500 mg or maximum tolerated dose (at least 1000mg daily), with or without insulin secretagogue (SU or glinides) or DPP-4 inhibitors or SGLT-2 inhibitors or alpha-glucosidase inhibitors for at least 8 weeks at a stable dose. The dose(s) of OAD other than metformin should be minimum half of the daily maximal dose according to local labelling or maximum tolerated dose.
* Insulin naïve. short-term insulin treatment (consecutive or cumulative treatment of ≤14 days) and insulin treatment for gestational diabetes are allowed.
* HbA1c 7.0-10.0 % (53-85 mmol/mol) (both inclusive)
* BMI 19-40 kg/m2 (both inclusive)

Exclusion Criteria:

* Known or suspected allergy or intolerance to the active substance or to any of the excipients of the investigational medical products
* Severe hypoglycemia during the previous 6 months.
* Hospitalization for diabetic ketoacidosis or hyperglycemic hyperosmolar syndrome during the previous 6 months.
* Cardiovascular disease within the last 12 months, defined as: stroke, decompensated heart failure (New York Heart Association [NYHA] class III or IV), myocardial infarction, or hospitalization for unstable angina pectoris or transient ischemic attack.
* Diagnosis of malignant neoplasms (except basal cell or squamous cell skin cancer, polyps and in-situ carcinomas) within the last 5 years or increased risk of cancer or relapse of cancer.
* Any antidiabetic medication other than permitted in the inclusion criteria or any weight-loss drug within the last 8 weeks..
* Systemic or intra-articular corticosteroids treatment within the last 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-05-28 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Week 0 to Week 16
  Change from baseline in Glycosylated Haemoglobin after 16 weeks of treatment

SECONDARY OUTCOMES:
Proportion of subjects reaching HbA1c targets | Week 0 to Week 16
  HbA1c <7% or HbA1c ≤6.5%
Change in FPG | Week 0 to Week 16
  Change from baseline in FPG after 16 weeks of treatment
9-point SMPG profiles | Week 0 to Week 16
  Mean plasma glucose, Postprandial and nocturnal increments, Fluctuation of 9-point SMPG. Plasma glucose measured: before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner,120 minutes after start of dinner, before bedtime, at 4 am and before breakfast.
Pre-breakfast SMPG | Week 0 to Week 16
  Mean plasma glucose, Within-subject variability of pre-breakfast SMPG.
Titration target | Week 0 to Week 16
  Proportion of subjects and time reaching titration targets
Numbers of hypoglycaemic episodes according to 2017 ADA/EASD classfication | Week 0 to Week 16
  Classification of hypoglycaemia: Level 1(glucose level below 3.9 mmol/L), Level 2(glucose level below 3.0 mmol/L) and Level 3(Severe hypoglycemia, denotes severe cognitive impairment requiring external assistance for recovery).
Numbers of injection site reactions | Week 0 to Week 16
  The injection site reactions was assessed during the treatment period of 16 weeks.
Frequency and severity of adverse events | Week 0 to Week 16 + 14 days follow-up
  Severity assessed by investigator. Mild: no or transient symptoms, no interference with subject's daily activities, no or minimal medical treatment. Moderate: marked symptoms, interference with subject's daily activities，and medical treatment for alleviation without grave or permanent injury to the subject. . Severe: considerable interference with subject's daily activities， and intensive treatment and intervention needed.
Anti-drug Antibodies: Anti-INS068 Antibodies | Week 0 to Week 16+14 days follow-up
  Number of Participants Positive or Negative for Anti-INS068 Antibodies were reported.
Changes in Body Weight | Week 0 to Week 16
  Change of body weight was evaluated from Week 0 to Week 16
Changes in Body Mass Index | Week 0 to Week 16
  Change of Body Mass Index was evaluated from Week 0 to Week 16
Change in Health Related Quality of Life Questionnaire (SF -36) | Week 0 to Week 16
  Change from baseline in scores of Health-Related Quality of Life Questionnaire after 16 weeks of treatment. The questionnaire contains 36 items across 8 domains and 2 summary scores. Score range: 0 (worst score) to 100 (best score)
Serum INS068 concentration | Week 0 to Week 16
  To evaluate PK of INS068

CONTACTS AND LOCATIONS:
Locations (35):
- United States (15):
  - National Research Institute - Huntington Park, Huntington Park, California
  - Clinical Trials Research, Lincoln, California
  - Torrance Clinical Research Institute Inc, Lomita, California
  - National Research Institute - Wilshire, Los Angeles, California
  - ALL Medical Research, LLC, Cooper City, Florida
  - New Generation of Medical Research, Hialeah, Florida
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Endocrinology Associates, Inc, Columbus, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Juno Research, LL, Houston, Texas
  - Juno Research, LLC - Medical Center Office, Houston, Texas
  - Juno Research, LLC - Southwest Houston Site, Houston, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
- Australia (3):
  - Core Research Group Pty Ltd, Brisbane, Queensland
  - The Royal Melbourne Hospital, Melbourne, Victoria
  - Austin Health (Heidelberg Repatriation Hospital), Melbourne, Victoria
- China (17):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Hainan General Hospital, Haikou, Hainan
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College, Huazhong University of Scince and Technology, Wuhan, Hubei
  - Nanjing Drum Tower Hospital,The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Zhongda Hospital Affiliated to Southeast University, Nanjing, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Shengjing Hospital Of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shanghai Xuhui District Central Hospital, Shanghai, Shanghai Municipality
  - Shanghai Putuo District Central Hospital, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan